CLINICAL TRIAL: NCT00187265
Title: Triple Resynchronization in Paced Heart Failure Patients
Brief Title: Trip HF Study: Triple Resynchronization in Paced Heeart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR03005HF
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Ventricular Dyssynchrony
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy

SUMMARY:
The purpose of this study is to evaluate the feasibility of permanent biventricular pacing using three ventricular leads, and its efficacy in terms of inter and intra-ventricular resynchronization, in patients with congestive heart failure and a non-functional atrium (chronic AF).

ELIGIBILITY:
Inclusion Criteria:

• NYHA class III-IV congestive heart failure, in spite of optimal medical treatment for their congestive heart failure for 1 month.

The medical treatment must include a 40 mg/day minimum dose of furosemide (or equivalent);

* Permanent atrial fibrillation (AF);
* Left ventricular ejection fraction (LVEF) ≤ 35%;
* Indication for a pacemaker implantation for a permanent and symptomatic bradycardia, or already implanted pacemaker under the condition that leads positioning corresponds to the criteria described in the protocol;
* Aortic pre-ejection delay at least equal to 140 ms.

Exclusion Criteria:

* Indication for a cardiac defibrillator;
* Having presented a myocardial infarct within the previous 3 months;
* Having undergone cardiac surgery or coronary revascularization procedure within the previous 3 months, or being scheduled for such procedures;
* Presenting chronic pulmonary insufficiency;
* Patients whose congestive heart failure requires the use of an intravenous inotropic support;
* Presenting a dysthyreosis;
* Having a life expectancy of less than one year, for other reasons than the congestive heart failure;
* Unable to be followed-up in the scope of the study for geographical reasons;
* Having refused to give their consent;
* Minors (age < 18 years) and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Study Completion 2005-10

PRIMARY OUTCOMES:
Z-ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Daubert, Principal Investigator — CHU Pontchaillou Rennes France
Locations (1):
- Department of Cardiology - CHU Pontchaillou, Rennes, France